CLINICAL TRIAL: NCT01639339
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Belimumab Plus Standard of Care Versus Placebo Plus Standard of Care in Adult Subjects With Active Lupus Nephritis
Brief Title: Efficacy and Safety of Belimumab in Patients With Active Lupus Nephritis
Acronym: BLISS-LN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114054; 2011-004570-28 (EudraCT Number)
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Lupus Nephritis
Keywords: Antibodies; Systemic Lupus Erythematosus; Autoimmune Disease; Glomerulonephritis; Belimumab; Lupus; Nephritis; Kidney Diseases; SLE
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic; Autoimmune Diseases; Glomerulonephritis; Nephritis; Kidney Diseases | interventions — Standard of Care; belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo plus standard therapy (Placebo Comparator): Placebo IV plus standard therapy; placebo administered on Days 0, 14, 28, and then every 28 days thereafter through Week 100, with a final evaluation at Week 104 in the double-blind period. In the open-label extension period, placebo patients who opt to participate will receive belimumab 10 mg/kg IV every 28 days for an additional 6 months.
  Interventions: Biological: Placebo plus standard therapy; Drug: Standard therapy
- Belimumab 10 mg/kg plus standard therapy (Experimental): Belimumab 10 mg/kg IV plus standard therapy; belimumab administered on Days 0, 14, 28, and then every 28 days thereafter through Week 100, with a final evaluation at Week 104 in the double-blind period. In the open-label extension period, patients who opt to participate will continue to receive belimumab 10 mg/kg IV every 28 days for an additional 6 months.
  Interventions: Biological: Belimumab 10 mg/kg plus standard therapy; Drug: Standard therapy

INTERVENTIONS:
Biological: Placebo plus standard therapy — Placebo plus standard therapy
  Arms: Placebo plus standard therapy
Biological: Belimumab 10 mg/kg plus standard therapy — Belimumab 10 mg/kg plus standard therapy
  Other Names: BENLYSTA™
  Arms: Belimumab 10 mg/kg plus standard therapy
Drug: Standard therapy — The standard therapies allowed in this study are:
  - High-dose steroids (for example, methylprednisolone) plus cyclophosphamide for induction therapy followed by azathioprine for maintenance therapy
  OR
  - High-dose steroids plus mycophenolate for induction therapy followed by mycophenolate for maintenance therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of belimumab in adult patients with active lupus nephritis.

DETAILED DESCRIPTION:
Study participants receive standard therapy (induction and maintenance) for lupus nephritis in addition to receiving either placebo (no active medicine) or belimumab. Induction therapy starts before the first dose of study drug (belimumab or placebo). Maintenance therapy begins after completion of induction therapy and continues for the remainder of the study. Participants receive study drug throughout the entire study, during both induction and maintenance periods. The controlled period of the study is 104 weeks. The random assignment in this study is "1 to 1" which means you have an equal chance of receiving treatment with belimumab or placebo. Participants who successfully complete the 104-week study may enter into a 6-month open-label extension. All participants in the open-label extension receive belimumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria.
* Biopsy confirmed active lupus nephritis.
* Clinically active lupus renal disease at screening requiring /receiving induction therapy with Standard of Care medications.
* Autoantibody-positive.

Key Exclusion Criteria:

* Pregnant or nursing.
* On dialysis within the past year.
* Treatment with belimumab within the past year .
* Receipt of induction therapy with cyclophosphamide within 3 months prior to induction therapy for the study.
* Receipt of any B cell targeted therapy (for example, rituximab), investigational biological agent within the past year.
* Severe active central nervous system (CNS) lupus.
* Required management of acute or chronic infections within the past 60 days.
* Current drug or alcohol abuse or dependence.
* Tested positive for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* History of severe allergic reaction to contrast agents or biological medicines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (106):
- United States (16):
  - GSK Investigational Site, La Palma, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Onalaska, Wisconsin
- Argentina (6):
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mendoza
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Brazil (8):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Juiz de Fora, Minas Gerais
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Goiânia
  - GSK Investigational Site, Lajeado
  - GSK Investigational Site, Salvador
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Montreal, Quebec
- China (13):
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Nanning
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Xi'an
- GSK Investigational Site, Bogotá, Colombia
- Czechia (2):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- France (7):
  - GSK Investigational Site, Cean Cedex 09
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (10):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Göttingen
- GSK Investigational Site, Hong Kong, Hong Kong
- Hungary (2):
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Szeged
- Mexico (5):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, México
  - GSK Investigational Site, México, D.F.
- Netherlands (3):
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Maastricht
- Philippines (5):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Lipa City, Batangas
  - GSK Investigational Site, Manila
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ufa
- South Korea (7):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Jeju Special Self-Governing Prov.
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo/ Pontevedra
- Taiwan (3):
  - GSK Investigational Site, Gueishan Township,Taoyuan County
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
- Thailand (4):
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Muang
  - GSK Investigational Site, Rajathevee
  - GSK Investigational Site, Saimai
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Anders HJ, Furie R, Malvar A, Zhao MH, Hiromura K, Weinmann-Menke J, Green Y, Jones-Leone A, Negrini D, Levy RA, Lightstone L, Tanaka Y, Rovin BH. Effect of belimumab on kidney-related outcomes in patients with lupus nephritis: post hoc subgroup analyses of the phase 3 BLISS-LN trial. Nephrol Dial Transplant. 2023 Nov 30;38(12):2733-2742. doi: 10.1093/ndt/gfad167. PMID 37463054
- [Derived] Sada K, Kurita N, Noma H, Matsuki T, Quasny H, Levy RA, Jones-Leone AR, Gairy K, Yajima N. MOONLIGHT study: the design of a comparative study of the effectiveness of belimumab in patients with a history of lupus nephritis from the post-Marketed effectiveness of belimumab cOhOrt and JapaN Lupus NatIonwide reGistry (LUNA) coHorT. Lupus Sci Med. 2022 Sep;9(1):e000746. doi: 10.1136/lupus-2022-000746. PMID 37017254
- [Derived] Furie R, Rovin BH, Houssiau F, Contreras G, Teng YKO, Curtis P, Green Y, Okily M, Madan A, Roth DA. Safety and Efficacy of Belimumab in Patients with Lupus Nephritis: Open-Label Extension of BLISS-LN Study. Clin J Am Soc Nephrol. 2022 Nov;17(11):1620-1630. doi: 10.2215/CJN.02520322. Epub 2022 Oct 27. PMID 36302567
- [Derived] Yu X, Chen N, Xue J, Mok CC, Bae SC, Peng X, Chen W, Ren H, Li X, Noppakun K, Gilbride JA, Green Y, Ji B, Liu C, Madan A, Okily M, Tang CH, Roth DA. Efficacy and Safety of Belimumab in Patients With Lupus Nephritis: Subgroup Analyses of a Phase 3 Randomized Trial in the East Asian Population. Am J Kidney Dis. 2023 Mar;81(3):294-306.e1. doi: 10.1053/j.ajkd.2022.06.013. Epub 2022 Sep 2. PMID 36058429
- [Derived] Rovin BH, Furie R, Teng YKO, Contreras G, Malvar A, Yu X, Ji B, Green Y, Gonzalez-Rivera T, Bass D, Gilbride J, Tang CH, Roth DA. A secondary analysis of the Belimumab International Study in Lupus Nephritis trial examined effects of belimumab on kidney outcomes and preservation of kidney function in patients with lupus nephritis. Kidney Int. 2022 Feb;101(2):403-413. doi: 10.1016/j.kint.2021.08.027. Epub 2021 Sep 22. PMID 34560137
- [Derived] Furie R, Rovin BH, Houssiau F, Malvar A, Teng YKO, Contreras G, Amoura Z, Yu X, Mok CC, Santiago MB, Saxena A, Green Y, Ji B, Kleoudis C, Burriss SW, Barnett C, Roth DA. Two-Year, Randomized, Controlled Trial of Belimumab in Lupus Nephritis. N Engl J Med. 2020 Sep 17;383(12):1117-1128. doi: 10.1056/NEJMoa2001180. PMID 32937045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated safety and efficacy of intravenous (IV) belimumab 10 mg/kg plus standard of care (SoC) compared to placebo plus SoC in adult participants with active lupus nephritis. This was a Phase 3, multi-center, multi-national study consisting of a randomized, double-blind, placebo-controlled period and an open-label extension period. The study was conducted in 21 countries.
Pre-assignment Details: A total of 797 participants were screened of which 349 participants failed screening and 448 participants were randomized in double-blind period. In open-label period, a total of 257 participants were enrolled of which 2 participants did not receive open-label study treatment and 255 participants received open-label belimumab.
Groups:
- Placebo to Belimumab 10 mg/kg: Participants were randomized to receive matching placebo intravenous (IV) plus standard of care (SoC) on Days 0 (Baseline), 14, 28 and then every 28 days thereafter through 100 Weeks with a final evaluation for the double-blind treatment period at Week 104. The randomization was stratified by their induction regimen (high dose cortiocsteroids [HDCS] plus Cyclophosphamide [CYC] versus [vs.] HDCS plus Mycophenolate Mofetil [MMF]) and race. After completing the double-blind period, eligible participants that were randomized to placebo IV plus SOC received Belimumab 10 milligram per kilogram (mg/kg) every 28 days until Week 24 with a final evaluation at Week 28 (4 weeks after the last dose) in open-label extension period.
- Belimumab 10 mg/kg to Belimumab 10: Participants were randomized to receive Belimumab 10 mg/kg IV plus SoC on Days 0 (Baseline), 14, 28 and then every 28 days thereafter through 100 Weeks with a final evaluation for the double-blind treatment period at Week 104. The randomization was stratified by their induction regimen (HDCS plus CYC vs. HDCS plus MMF) and race. After completing the double-blind period, eligible participants that were randomized to belimumab 10 mg/kg IV plus SOC continued to receive Belimumab 10 mg/kg every 28 days until Week 24 with a final evaluation at Week 28 (4 weeks after the last dose) in open-label extension period.
Period: Double-blind Period (Up to Week 104)
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10
Started | 224 | 224
Completed | 170 | 186
Not Completed | 54 | 38
Not completed — Withdrawal by Subject | 26 | 19
Not completed — Physician Decision | 11 | 5
Not completed — Lost to Follow-up | 5 | 4
Not completed — Protocol Violation | 0 | 2
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse Event | 10 | 7
Period: Open-label Period (Up to Week 28)
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10
Started | 123 (Of the 356 participants who completed the double-blind period, 279 were eligible for open-label treatment. As enrolling into the open-label period was optional, only 257 participants enrolled, of whom 255 started open-label treatment.) | 132
Completed | 122 | 124
Not Completed | 1 | 8
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10 | Total
Number analyzed (Participants) | 224 | 224 | 448
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (10.64) | 33.7 (10.73) | 33.4 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 198 | 394
  Male | 28 | 26 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian (AI) or Alaska Native (AN) | 6 | 4 | 10
  Asian-Central/South Asian Heritage (H) | 2 | 3 | 5
  Asian-Japanese/East Asian/Southeast Asian H | 107 | 112 | 219
  Mixed Asian | 1 | 0 | 1
  Black or African American (AA) | 31 | 30 | 61
  White/Caucasian/European H | 71 | 72 | 143
  White/Caucasian/Arabic/North African H | 4 | 1 | 5
  Multiple-AA/African H and AI or AN and White | 1 | 1 | 2
  Multiple-Asian and White | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Period: Percentage of Participants With Primary Efficacy Renal Response (PERR) at Week 104
Description: PERR is defined as urinary protein creatinine ratio <=0.7, estimated glomerular filtration rate (eGRF) was not more than 20 percent (%) below the pre-flare value or >=60 milliliters per minute per 1.73 square meter (mL/min/1.73m^2) and was not a treatment failure. Analysis was performed using a logistic regression model for the comparison between Belimumab and Placebo with covariates treatment group, induction regimen (CYC vs. MMF), race (Black vs. Non-Black), Baseline urine protein-creatinine ratio (uPCR), and Baseline eGFR. Modified Intent-to-treat (mITT) Population consisted of all randomized participants who received at least one dose of study treatment and were not excluded due to Good Clinical Practice (GCP) non-compliance. Percentage of participants with PERR at Week 104 has been presented.
Time Frame: Week 104
Population: mITT Population.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Participants were randomized to receive matching placebo IV plus SoC on Days 0 (Baseline), 14, 28 and then every 28 days thereafter through 100 Weeks with a final evaluation for the double-blind treatment period at Week 104. The randomization was stratified by their induction regimen (high dose cortiocsteroids [HDCS] plus Cyclophosphamide [CYC] versus [vs.] HDCS plus Mycophenolate Mofetil [MMF]) and race.
- Belimumab 10 mg/kg: Participants were randomized to receive Belimumab 10 milligrams per kilogram (mg/kg) IV plus SoC on Days 0 (Baseline), 14, 28 and then every 28 days thereafter through 100 Weeks with a final evaluation for the double-blind treatment period at Week 104. The randomization was stratified by their induction regimen (HDCS plus CYC vs. HDCS plus MMF) and race.
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 223 | 223
Percentage of participants | 32.3 | 43.0
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; p = 0.0311, Regression, Logistic — P-value was calculated using logistic regression model. Test 1 of 5 in a step-down sequential testing procedure; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.04 to 2.32] — Treatment comparison between Belimumab 10 mg/kg and placebo using odds ratio and its corresponding 95% confidence interval has been presented

2. Secondary Outcome: Double-blind Period: Percentage of Participants With Complete Renal Response (CRR) at Week 104
Description: CRR is defined as urinary protein creatinine ratio <0.5, eGRF was not more than 10% below the pre-flare value or >=90 mL/min/1.73m^2 and was not a treatment failure. Analysis was performed using a logistic regression model for the comparison between Belimumab and Placebo with covariates of induction regimen (CYC vs. MMF), race (Black vs. Non-Black), Baseline uPCR and Baseline eGFR. Percentage of participants with CRR at Week 104 has been presented.
Time Frame: Week 104
Population: mITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 223 | 223
Percentage of participants | 19.7 | 30.0
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; p = 0.0167, Regression, Logistic — P-value was calculated using logistic regression model. Test 2 of 5 in a step-down sequential testing procedure; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.11 to 2.74] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Double-blind Period: Percentage of Participants With PERR at Week 52
Description: PERR is defined as urinary protein creatinine ratio <=0.7, eGRF was not more than 20% below the pre-flare value or >=60 mL/min/1.73m^2 and was not a treatment failure. Analysis was performed using a logistic regression model for the comparison between Belimumab and Placebo with covariates of induction regimen (CYC vs. MMF), race (Black vs. Non-Black), uPCR, and Baseline eGFR. Percentage of participants with PERR at Week 52 has been presented.
Time Frame: Week 52
Population: mITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 223 | 223
Percentage of participants | 35.4 | 46.6
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; p = 0.0245, Regression, Logistic — P-value was calculated using logistic regression model. Test 3 of 5 in a step-down sequential testing procedure; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.06 to 2.38] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Double-blind Period: Number of Participants With Time to Death or Renal Related Event
Description: Events are defined as the first event experienced among the following: death, progression to end stage renal disease, doubling of serum creatinine from Baseline, renal worsening or renal-related treatment failure. Participants who discontinued randomized treatment, withdrew from the study, were lost to follow-up, or had a non renal-related treatment failure were censored. Participants who completed the 104-week treatment period were censored at the Week 104 visit. Time to event is defined as event date minus treatment start date plus one. Analysis was performed using Cox proportional hazards model for the comparison between Belimumab and Placebo adjusting for induction regimen, race, Baseline uPCR and Baseline eGFR. Number of participants with time to death or renal related event up to Week 104 has been presented.
Time Frame: Up to Week 104
Population: mITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 223 | 223
Participants | 63 | 35
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; p = 0.0014, Cox proportional hazards model — P-value was calculated using Cox proportional hazards model. Test 4 of 5 in a step-down sequential testing procedure; Cox Proportional Hazard = 0.51, 95% CI 2-sided [0.34 to 0.77] — Treatment comparison between Belimumab 10 mg/kg and placebo using Cox proportional hazards ratio and its corresponding 95% confidence interval has been presented

5. Secondary Outcome: Double-blind Period: Percentage of Participants With Ordinal Renal Response (ORR) at Week 104
Description: ORR is defined with respect to reproducible responses that included CRR, partial RR (PRR) and non responder. CRR is reported when uPCR was <0.5, eGFR was not more than 10% below pre-flare GFR or within normal range and not a treatment failure. PRR is >=50% decrease from Baseline in uPCR and one of the following: value <1 if Baseline <=3, or value <3 if the Baseline was >3, eGFR not more than 10% below Baseline GFR or within normal range and not a treatment failure and not a CRR. Non responder is reported when neither CRR nor PRR criteria was met. Percentage of participants reporting CRR, PRR and non responders at Week 104 has been presented.
Time Frame: Week 104
Population: mITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 223 | 223
Percentage of participants
  CRR | 19.7 | 30.0
  PRR | 17.0 | 17.5
  Non responder | 63.2 | 52.5
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Other; p = 0.0096, Rank ANCOVA — P-value is rank analysis of covariance model comparing Belimumab and Placebo with covariates for treatment group, induction regimen(CYC vs MMF),race(Black vs Non-black), Baseline uPCR, and eGFR. Test 5 of 5 in step-down sequential testing procedure

6. Secondary Outcome: Double-blind Period: Number of Participants Reporting On-treatment AEs and SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is any untoward medical occurrence that, at any dose: resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Number of participants with on-treatment AEs and SAEs has been reported.
Time Frame: Up to Week 104
Population: Safety Population comprised of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 224 | 224
Participants
  Any AE | 211 | 214
  Any SAE | 67 | 58

7. Secondary Outcome: Double-blind Period: Number of Participants Reporting AESI
Description: An AESI is one of scientific and medical concern specific to the product, for which ongoing monitoring and rapid communication by investigator to sponsor can be appropriate. A summary of protocol defined AESIs include malignant neoplasms including and excluding non-melanoma skin cancer (NMSC), post-infusion systemic reactions (PISR), all infections of special interest (opportunistic infections [OI], Herpes Zoster [HZ], tuberculosis [TB], and sepsis), depression (including mood disorders and anxiety)/suicide/self-injury and deaths. On-treatment data is displayed.
Time Frame: Up to Week 104
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Belimumab 10 mg/kg
Number analyzed (Participants) | 224 | 224
Participants
  Malignancies excluding NMSC | 0 | 2
  Malignancies including NMSC | 0 | 3
  PISR | 29 | 26
  All infections of special interest | 34 | 30
  Depression/suicide/self-injury | 16 | 11
  Deaths | 3 | 4

8. Primary Outcome: Open-label Period: Number of Participants Reporting Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is any untoward medical occurrence that, at any dose: resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Number of participants with AEs and SAEs have been reported.
Time Frame: From first open-label dose (Day 1) up to open-label Week 32 (8 weeks after last dose)
Population: Safety Open-Label Population comprised of all participants who received at least one dose of open-label treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Belimumab 10 mg/kg to Belimumab 10 mg/kg: Participants were randomized to receive Belimumab 10 mg/kg IV plus SoC on Days 0 (Baseline), 14, 28 and then every 28 days thereafter through 100 Weeks with a final evaluation for the double-blind treatment period at Week 104. The randomization was stratified by their induction regimen (HDCS plus CYC vs. HDCS plus MMF) and race. After completing the double-blind period, eligible participants that were randomized to belimumab 10 mg/kg IV plus SOC continued to receive Belimumab 10 mg/kg every 28 days until Week 24 with a final evaluation at Week 28 (4 weeks after the last dose) in open-label extension period.
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10 mg/kg
Number analyzed (Participants) | 123 | 132
Participants
  Any AE | 76 | 92
  Any SAE | 5 | 10

9. Primary Outcome: Open-label Period: Number of Participants Reporting Adverse Events of Special Interest (AESI)
Description: An AESI is one of scientific and medical concern specific to the product, for which ongoing monitoring and rapid communication by investigator to sponsor can be appropriate. A summary of protocol defined AESIs include malignant neoplasms including and excluding non-melanoma skin cancer (NMSC), post-infusion systemic reactions (PISR), all infections of special interest (opportunistic infections [OI], Herpes Zoster [HZ], tuberculosis [TB], and sepsis), depression (including mood disorders and anxiety)/suicide/self-injury and deaths.
Time Frame: From first open-label dose (Day 1) up to open-label Week 32 (8 weeks after last dose)
Population: Safety Open-Label Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10 mg/kg
Number analyzed (Participants) | 123 | 132
Participants
  Malignancies excluding NMSC | 0 | 0
  Malignancies including NMSC | 0 | 0
  PISR | 4 | 5
  All infections of special interest | 2 | 6
  Depression/suicide/self-injury | 2 | 4
  Deaths | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-SAEs and SAEs were summarised from the start of the first treatment up to Week 104 in double-blind period and from the first open-label dose up to Week 32 (8 weeks after last dose) in open-label extension period.
Description: All-cause mortality, non-SAEs and SAEs were reported for safety population (double-blind period) and safety open-label population (open-label period). Non-serious adverse events not meeting 5% in the open label period were reported as 0% incidence but could have incidences between 0 and 5%.
Arm/Group | Placebo | Belimumab 10 mg/kg | Placebo to Belimumab 10 mg/kg | Belimumab 10 mg/kg to Belimumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 5/224 | 6/224 | 1/123 | 0/132
Serious Adverse Events (participants affected / at risk) | 78/224 | 65/224 | 5/123 | 10/132
Other Adverse Events (participants affected / at risk) | 191/224 | 186/224 | 34/123 | 39/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=224) | Belimumab 10 mg/kg (N=224) | Placebo to Belimumab 10 mg/kg (N=123) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (N=132)
Pneumonia (Infections and infestations) | 10 (11) | 10 (11) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes oesophagitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary nocardiosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhodococcus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 8 (10) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serositis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Central nervous system lupus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis uraemic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal biophysical profile score equivocal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunosuppression (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=224) | Belimumab 10 mg/kg (N=224) | Placebo to Belimumab 10 mg/kg (N=123) | Belimumab 10 mg/kg to Belimumab 10 mg/kg (N=132)
Upper respiratory tract infection (Infections and infestations) | 74 (134) | 81 (159) | 14 (18) | 23 (24)
Urinary tract infection (Infections and infestations) | 37 (72) | 43 (73) | 10 (12) | 12 (14)
Nasopharyngitis (Infections and infestations) | 31 (50) | 35 (60) | 8 (9) | 3 (3)
Gastroenteritis (Infections and infestations) | 23 (28) | 21 (24) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 19 (26) | 18 (24) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 19 (20) | 17 (17) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 5 (5) | 13 (13) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 48 (56) | 45 (59) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 24 (33) | 21 (28) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (21) | 16 (25) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 12 (15) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 15 (18) | 9 (10) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 16 (16) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (52) | 26 (44) | 5 (5) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 17 (24) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 (18) | 18 (25) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 12 (14) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 35 (57) | 34 (51) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 19 (21) | 13 (18) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 13 (17) | 16 (23) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 17 (20) | 11 (14) | 0 (0) | 0 (0)
Fatigue (General disorders) | 14 (15) | 12 (12) | 0 (0) | 0 (0)
Oedema (General disorders) | 12 (15) | 9 (9) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 23 (26) | 13 (16) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 19 (29) | 15 (28) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 17 (18) | 23 (31) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 9 (11) | 12 (13) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 30 (38) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (23) | 24 (36) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 20 (23) | 12 (14) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 18 (19) | 10 (10) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT01639339/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT01639339/SAP_002.pdf